CLINICAL TRIAL: NCT06154538
Title: Comparison of Immune Checkpint Inhibitors Combined With Chemotherapy Versus Chemotherapy Alone in the Neoadjuvant Treatment of Locally Advanced Colorectal Cancer: a Randomized, Open-label, Single-center Phase II Clinical Study
Brief Title: Immune Checkpoint Inhibitors + Chemotherapy Versus Chemotherapy in the Neoadjuvant Treatment of Locally Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, QIAN LIU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS-NCTplusAK104
Record Dates: First submitted 2023-11-12; First posted 2023-12-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Colorectal Carcinoma
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICIs + FOLFOX group (Experimental): Patients in this group will receive ICIs combined with FOLFOX regimen, specifically: ICIs, intravenous infusion, D1; Oxaliplatin (85mg/m2), intravenous infusion, D1; Calcium folinate (400mg/m2), intravenous infusion, D1; 5-FU (400mg/m2), intravenous infusion, D1, then continuous intravenous infusion of 1200mg/(m2·d)×2d (total amount of 2400mg/m2, infusion for 46-48h) every two weeks. Imaging evaluation will be performed after 3 cycles of preoperative treatment. If the disease is resectable, surgery will be performed. If R0 resection is achieved, the preoperative regimen will continue for up to 9 cycles.
  Interventions: Drug: Immune checkpoint inhibitor; Drug: FOLFOX regimen
- FOLFOX group (Active Comparator): Patients in this group will undergo FOLFOX chemotherapy regimen, specifically: Oxaliplatin 85 mg/m2 dissolved in 500 ml of 5% glucose solution, intravenous drip, on Day 1, in combination with calcium folinate (400mg/m2), intravenous infusion, on Day 1, and 5-FU (400mg/m2), intravenous infusion, on Day 1, followed by continuous intravenous infusion of 1200mg/(m2·d) for 2 days (total dose of 2400mg/m2, infusion for 46-48 hours), once every 2 weeks. After 3 cycles of preoperative treatment, imaging evaluation will be performed. If the disease is resectable, surgery will be performed. If R0 resection is achieved, the preoperative treatment regimen will be continued after surgery, for a maximum of 9 cycles.
  Interventions: Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — PD-1 antibody
  Other Names: 1
  Arms: ICIs + FOLFOX group
Drug: FOLFOX regimen — FOLFOX chemotherapy
  Other Names: 0

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of the combination of immune checkpoint inhibitors (ICIs) and FOLFOX regimen compared to FOLFOX regimen alone in the neoadjuvant chemotherapy of locally advanced colorectal cancer. The main question aims to answer are:

Question 1: Compare the pathological complete response rate between the combination of ICIs and FOLFOX regimen and the FOLFOX alone.

Question 2: Compare the survival outcomes and safety between the combination of ICIs and FOLFOX regimen and the FOLFOX alone.

Two groups of participants will receive different new adjuvant chemotherapy regimens, and their efficacy will be compared.

DETAILED DESCRIPTION:
A prospective, randomized, open, multi-center clinical study evaluating the efficacy (pathological response, survival outcomes) and safety of the combination of ICIs and FOLFOX regimen compared to FOLFOX regimen in the treatment of locally advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75, no gender restrictions;
* Histologically or cytologically confirmed colorectal adenocarcinoma;
* Clinically diagnosed as stage II/III colorectal cancer based on CT and/or MRI (according to the 8th edition of AJCC staging);
* Sufficient tumor tissue specimens for mismatch repair protein expression or microsatellite instability testing;
* No prior systemic drug therapy and/or radiotherapy for colorectal adenocarcinoma;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Normal major organ function, no severe blood, heart, lung, liver, kidney dysfunction, or immune deficiency diseases (see protocol for details);
* Voluntary participation in this study and signed informed consent form;
* Expected good compliance to complete the study treatment, follow-up for efficacy and adverse reactions according to the protocol requirements.

Exclusion Criteria:

* Pathology is other malignant tumors besides adenocarcinoma, such as squamous cell carcinoma, gastrointestinal stromal tumor, melanoma, etc.;
* Within 5 years prior to the first use of investigational drug, diagnosed with other malignant tumors, excluding effectively treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or in situ cervical cancer and/or breast cancer effectively removed;
* Any distant metastatic colorectal adenocarcinoma (according to AJCC 8th edition staging, determined as M1), including but not limited to distant lymph node metastasis, liver metastasis, lung metastasis, intraperitoneal dissemination, or malignant peritoneal effusion;
* Various severe underlying diseases and autoimmune diseases (see protocol for details);
* Unable to control recurrent bleeding or subjects who received blood transfusion within 2 weeks prior to the first use of investigational drug;
* Any other circumstances where the investigator believes it may increase the risk associated with participating in the study, the administration of the investigational drug, or affect the subject's ability to receive the investigational drug and the reliability of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | at time of surgery
  pathological complete response rate

SECONDARY OUTCOMES:
R0 resection rate | at time of surgical assessment (after 3 cycles), up to 12 months
  R0 resection rate
DFS | up to 3 years after intervention
  disease-free survival
3 years DFS rate | 3 years
  3 years DFS rate
OS | at 1,2,3 years at follow-up time
  overall survival

OTHER OUTCOMES:
adverse event adverse event rate | 90 days
  adverse event
treatment-related adverse event | 90 days
  treatment-related adverse event
serious adverse event | 90 days
  serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Qian Liu, Principal Investigator — vice director of colorectal surgery dept.; Jing Huang, Study Director — vice director of medical oncology dept.
Locations (3):
- China (3):
  - Cancer Hospital/ National Cancer Center, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No